CLINICAL TRIAL: NCT04225923
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of NPC-21 for Kidney Transplant Recipients at High-Risk of Cytomegalovirus Infection
Brief Title: A Study for Kidney Transplant Recipients at High-Risk of Cytomegalovirus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NPC-21-2
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cytomegalovirus Disease
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NPC-21 Low dose (Experimental): NPC-21 (6mg/kg) will be administered
  Interventions: Drug: NPC-21 Low dose
- NPC-21 High dose (Experimental): NPC-21 (12mg/kg) will be administered
  Interventions: Drug: NPC-21 High dose
- NPC-21 Placebo (Placebo Comparator): Placebo (normal saline) will be administered
  Interventions: Drug: NPC-21 Placebo

INTERVENTIONS:
Drug: NPC-21 Low dose — NPC-21 will be administered via an approximately 60-minute intravenous infusion on Day 1 and at Week 4, 8, 12
  Arms: NPC-21 Low dose
Drug: NPC-21 High dose — NPC-21 will be administered via an approximately 60-minute intravenous infusion on Day 1 and at Week 4, 8, 12
  Arms: NPC-21 High dose
Drug: NPC-21 Placebo — Placebo will be administered via an approximately 60-minute intravenous infusion on Day 1 and at Week 4, 8, 12
  Arms: NPC-21 Placebo

SUMMARY:
The primary objective is to assess the efficacy and safety of NPC-21 when administered prophylactically to cytomegalovirus (CMV) seronegative patients receiving a first kidney transplant from a CMV seropositive donor.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled study of NPC-21 for kidney transplant recipients at high risk of CMV infection in the United States and Japan. Approximately 108 eligible patients will be randomized prior to first study drug administration to receive low-dose NPC 21, high-dose NPC-21, or placebo. Randomization will be stratified by region (United States or Japan)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 to 75 years of age in the United States or 20 to 75 years of age in Japan at the time of obtaining informed consent.
2. Patients must be CMV seronegative pre-transplant and scheduled to receive or have received (within 7 days prior to first study drug administration) a first kidney transplant from a CMV seropositive donor.
3. Patients must be willing and able to give written informed consent for participation in the study.
4. Patients must be eligible to undergo kidney transplantation from a living or deceased donor, as per institutional standards.
5. Patients must agree with contraception by using appropriate contraceptive measures.

Exclusion Criteria:

1. Patients who have received a previous solid organ transplantation or hematopoietic stem cell transplantation.
2. Patients who receive a multi-organ transplant.
3. Patients who have CMV disease or CMV viremia at Screening.
4. Patients who have a positive donor-specific antibody within 90 days prior to Randomization confirmed via medical records.
5. Patients whose body weight is more than 120 kg at Screening.
6. Patients who have received the following anti-CMV therapy within 7 days prior to Randomization and/or plan to receive the following anti-CMV therapy during the study:

   ・ Anti-CMV agents (eg, foscarnet, ganciclovir, valganciclovir, letermovir, high dose acyclovir, high dose valacyclovir, high dose famciclovir, or cidofovir).

   Note: The use of anti-CMV agents per local standard of care during the Rescue Phase of the study is permitted.

   Note: The use of anti-herpes simplex virus and anti-varicella zoster virus prophylaxis for at-risk patients is recommended (as long as the doses are below the one specified above).
7. Patients who have received the following therapy within 28 days prior to Randomization and/or plan to receive the following anti-CMV therapy during the study:

   * CMV hyperimmune globulin (eg, CytoGam).
   * Intravenous immunoglobulin.
   * Plasmapheresis (receipt prior to first study drug administration is acceptable).
8. Patients with a history of a serious drug allergy to proteins, immunoglobulins, transfusions, or vaccines or any excipient of the NPC-21 formulation.
9. Patients with severe hepatic insufficiency at Screening (eg, Child-Pugh Class C).
10. Patients with active and untreated hepatitis B virus or hepatitis C virus, as documented as part of the pre-transplant screening.
11. Patients with known human immunodeficiency virus infection, based on medical records serology.
12. Patients with any uncontrolled infection at Randomization or a history of serious and uncontrolled infection within 6 months prior to Randomization.
13. Patients who are pregnant or lactating.
14. Patients with a history of malignancy within 5 years prior to Randomization other than curatively treated in situ cervical carcinoma, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma.
15. Patients with a history of alcohol or drug abuse or dependence within 1 year prior to Randomization that, in the opinion of the Investigator, would preclude study participation.
16. Patients who have previously participated in this study or any other study involving NPC-21.
17. Patients who have previously participated or are currently participating in any study involving the administration of a CMV vaccine or another CMV investigational agent.
18. Patients who have participated in another interventional clinical study and received another investigational product (ie, not approved by the Food and Drug Administration in the United States or the Ministry of Health, Labour and Welfare in Japan) within 90 days before Randomization.
19. Patients who are unable or unwilling, in the opinion of the Investigator, to comply with the protocol.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (14):
  - Mayo Clinic - Scottsdale, Phoenix, Arizona
  - California Institute of Renal Research, La Mesa, California
  - Piedmont Healthcare, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Renal Disease Research Institute, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin
- Japan (14):
  - Research site_204, Nagakute, Aichi-ken
  - Research site_201, Nagoya, Aichi-ken
  - Research site_202, Toyoake, Aichi-ken
  - Research site_206, Kobe, Hyōgo
  - Research site_205, Nishinomiya, Hyōgo
  - Research site_217, Kawasaki-shi, Kanagawa
  - Research site_212, Kumamoto, Kumamoto
  - Research site_215, Tomigusuku-shi, Okinawa
  - Research site_211, Osaka, Osaka
  - Research site_214, Osaka, Osaka
  - Research site_216, Osaka, Osaka
  - Research site_208, Suita, Osaka
  - Research site_203, Shimotsuke, Tochigi
  - Research site_213, Hachioji-shi, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ichimaru N, Natori Y, Alloway RR, Wojciechowski D, Castillo Almeida NE, Futamura K, Watanabe T, Nakagawa K, Egawa H; LionHeart21 Study Group. Phase 2, Randomized, Double-blind, Placebo-controlled Study of Fiztasovimab (NPC-21) for Kidney Transplant Recipients at High Risk of Cytomegalovirus Infection (LionHeart21). Transplantation. 2025 Jun 1;109(6):985-993. doi: 10.1097/TP.0000000000005260. Epub 2025 May 18. PMID 40072882
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2020 to August 2022, adult CMV seronegative patients who received a first kidney transplant from CMV seropositive donors were enrolled in the study at 31 sites in the United States and Japan.
Groups:
- NPC-21 Low Dose: NPC-21 (6mg/kg) will be administered
  NPC-21 Low dose : NPC-21 will be administered via an approximately 60-minute intravenous infusion
- NPC-21 High Dose: NPC-21 (12mg/kg) will be administered
  NPC-21 High dose : NPC-21 will be administered via an approximately 60-minute intravenous infusion
- NPC-21 Placebo: Placebo (normal saline) will be administered
  NPC-21 Placebo: Placebo will be administered via an approximately 60-minute intravenous infusion
Period: Overall Study
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Started | 38 | 11 | 38
Completed | 33 | 10 | 33
Not Completed | 5 | 1 | 5
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — A subject completed the study but was reported incorrectly in the report form | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- NPC-21 Low Dose: NPC-21 (6mg/kg) will be administered
  NPC-21 Low dose: NPC-21 will be administered via an approximately 60-minute intravenous infusion
- NPC-21 High Dose: NPC-21 (12mg/kg) will be administered
  NPC-21 High dose: NPC-21 will be administered via an approximately 60-minute intravenous infusion
- Total: Total of all reporting groups
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo | Total
Number analyzed (Participants) | 38 | 11 | 38 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 9 | 31 | 74
  >=65 years | 4 | 2 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.45) | 50.5 (15.65) | 51.7 (14.04) | 51.0 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 15 | 34
  Male | 23 | 7 | 23 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 10 | 3 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 1 | 10 | 18
  White | 19 | 6 | 17 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 8 | 28 | 64
  Japan | 10 | 3 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Incidence of CMV Disease or CMV Viremia
Description: The proportion of patients with CMV disease (CMV syndrome or tissue-invasive CMV disease) or CMV viremia (defined as the detection of 250 IU/mL in plasma measured by PCR analysis in central laboratory or meets the local criteria for CMV viremia measured by PCR analysis or antigenemia testing) per total patients through 16 weeks from first study drug administration.
  The non-responders include all patients who develop CMV disease or CMV viremia and patients who discontinue from the study in the absence of CMV disease or CMV viremia.
Time Frame: 16 weeks
Population: All patients who received a kidney transplant from a living or deceased donor and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
Participants | 29 | 9 | 26

2. Secondary Outcome: Incidence of CMV Disease or CMV Viremia
Description: The proportion of patients with CMV disease or CMV viremia. The non-responders include all patients who develop CMV disease or CMV viremia and patients who discontinue from the study in the absence of CMV disease or CMV viremia.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
Participants | 29 | 9 | 26

3. Secondary Outcome: Incidence of CMV Disease
Description: The proportion of patients with CMV disease
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
Participants | 2 | 0 | 5

4. Secondary Outcome: Incidence of CMV Viremia
Description: The proportion of patients with CMV viremia.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
Participants | 22 | 8 | 17

5. Secondary Outcome: Time to Detectable CMV Disease or CMV Viremia
Description: The count and proportion of patients experiencing event and censored will be summarized by treatment group.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
weeks | 6.1 [5.0 to 9.3] | 6.3 [4.1 to 8.3] | 6.3 [5.1 to NA] — Insufficient number of patients with events

6. Secondary Outcome: Time to Detectable CMV Disease
Description: The count and proportion of patients experiencing event and censored will be summarized by treatment group.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
weeks | NA [NA to NA] — Insufficient number of patients with events | NA [NA to NA] — Insufficient number of patients with events | NA [NA to NA] — Insufficient number of patients with events

7. Secondary Outcome: Time to Detectable CMV Viremia
Description: The count and proportion of patients experiencing event and censored will be summarized by treatment group.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
Number analyzed (Participants) | 38 | 11 | 38
weeks | 6.1 [5.0 to NA] — Insufficient number of patients with events | 6.3 [4.1 to 8.3] | NA [5.7 to NA] — Insufficient number of patients with events

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Non-serious and serious Treatment Emergent Adverse Events were reported.
Arm/Group | NPC-21 Low Dose | NPC-21 High Dose | NPC-21 Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/11 | 0/38
Serious Adverse Events (participants affected / at risk) | 17/38 | 3/11 | 25/38
Other Adverse Events (participants affected / at risk) | 33/38 | 9/11 | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NPC-21 Low Dose (N=38) | NPC-21 High Dose (N=11) | NPC-21 Placebo (N=38)
Cytomegalovirus viraemia (Infections and infestations) | 3 | 2 | 3
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 3
Cytomegalovirus syndrome (Infections and infestations) | 1 | 0 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 2
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 2 | 0 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal effusion (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 5
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Impaired healing (General disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 2 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NPC-21 Low Dose (N=38) | NPC-21 High Dose (N=11) | NPC-21 Placebo (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 6
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 4
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 3 | 15
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 10
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 3
Vomiting (Gastrointestinal disorders) | 5 | 0 | 4
Asthenia (General disorders) | 1 | 0 | 3
Chills (General disorders) | 2 | 0 | 2
Fatigue (General disorders) | 3 | 2 | 8
Oedema peripheral (General disorders) | 7 | 1 | 4
Pyrexia (General disorders) | 4 | 1 | 3
Peripheral swelling (General disorders) | 0 | 1 | 3
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 4
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 6 | 3 | 6
Cytomegalovirus viraemia (Infections and infestations) | 19 | 7 | 12
Polyomavirus viraemia (Infections and infestations) | 2 | 1 | 3
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 0 | 3
Incision site pain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Scrotal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 1 | 0
Weight decreased (Investigations) | 4 | 0 | 4
White blood cell count decreased (Investigations) | 2 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Donor specific antibody present (Investigations) | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Osteodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 7
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 7
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 6 | 2 | 6
Anxiety (Psychiatric disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 3
Perinephric collection (Renal and urinary disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 3
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypotension (Vascular disorders) | 2 | 0 | 4
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 3

LIMITATIONS AND CAVEATS:
Patients who developed CMV disease or CMV viremia received rescue therapy and administration of NPC-21 or Placebo was discontinued.

Patients who completed rescue therapy withdrew early from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04225923/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04225923/SAP_001.pdf